CLINICAL TRIAL: NCT04986553
Title: A Multi-Center, Prospective Registry to Evaluate the Continued Safety and Performance of Clavicle Plates
Status: Withdrawn | Type: Observational
Why Stopped: The study was suspended and terminated.
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AIRR-0005
Record Dates: First submitted 2021-06-22; First posted 2021-08-03 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Clavicle Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- 50 subjects, male and female, at least 18 years of age: 50 subjects who are candidates for surgery using the Arthrex Clavicle Plate for treatment of clavicle fractures.
  Interventions: Device: Arthrex Clavicle Plates

INTERVENTIONS:
Device: Arthrex Clavicle Plates — Arthrex Clavicle Plate for treatment of clavicle fractures

SUMMARY:
The objective of the registry is to evaluate the continued safety and performance of Arthrex Clavicle Plates used to treat clavicle fractures.

DETAILED DESCRIPTION:
To assess safety, device-related adverse events will be reported and evaluated over the course of the study. To evaluate the performance imaging of the target area will be evaluated at three months postoperative. Additionally, patient-reported outcomes will be evaluated at three months postoperative, 6 months postoperative, and one year postoperative using the Visual Analogue Scale (VAS), Veterans Rand 12-Item Health Survey (VR-12), and American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES).

ELIGIBILITY:
Inclusion Criteria:

1. The subject requires surgery using the Arthrex Clavicle Plate for clavicle fracture.
2. The subject is 18 years of age or over.
3. The subject is not considered a vulnerable subject (i.e., child, pregnant, nursing, prisoner, or ward of the state).
4. Subject signed informed consent and is willing and able to comply with all study requirements

Exclusion Criteria:

1. Insufficient quantity or quality of bone.
2. Blood supply limitations and previous infections, which may retard healing.
3. Foreign-body sensitivity.
4. Any active infection or blood supply limitations.
5. Conditions that tend to limit the patient's ability or willingness to restrict activities or follow directions during the healing period.
6. Subjects that are skeletally immature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Arthrex Clavicle Plates are intended to be used in the general population for clavicle fractures.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
To assess a change in Visual Analogue Scale (VAS) survey | Preoperatively, 3 months, 6 months and 12 months postoperatively
  Patient reported pain scale 0-10 point scale (0 min,10 max)
To assess a change in Veterans Rand 12-Item Health Survey (VR-12) | Preoperatively, 3 months, 6 months and 12 months postoperatively
  Patient reported changes in general health and mental survey. Average score is 50 (negative answers bring scores down, positive answers bring scores up
To assess a change in American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) | Preoperatively, 3 months, 6 months and 12 months postoperatively
  ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. There is one pain scale worth 50 points and ten activities of daily living worth 50 points.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sierra Pacific Orthpaedic CenterMedical Group, Inc, Fresno, California
  - Panorama Orthopedics & Spine Center, PC, Golden, Colorado